CLINICAL TRIAL: NCT02984670
Title: Cognitive Behavior Therapy for Insomnia: Analysis of Components, Mediators and Moderators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Markus Jansson-Fröjmark, PhD., Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBT-I CMM
Record Dates: First submitted 2016-11-21; First posted 2016-12-07 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Cognitive therapy; Behavior therapy; Moderation; Mediation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Negotiating | interventions — Cognitive Behavioral Therapy; Behavior Therapy; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Behavior Therapy (Experimental)
  Interventions: Behavioral: Behavior Therapy
- Cognitive Therapy (Experimental)
  Interventions: Behavioral: Cognitive Therapy
- Waitlist (Other)
  Interventions: Behavioral: Waitlist.

INTERVENTIONS:
Behavioral: Cognitive Therapy — Cognitive Therapy involves challenging negative automatic thoughts about sleep and the use of behavioral experiments to challenge and test five cognitive processes (i.e., worry, dysfunctional thoughts, monitoring, safety behaviours, misperception) proposed to perpetuate insomnia.
  Arms: Cognitive Therapy
Behavioral: Behavior Therapy — Behavior Therapy involves the use of stimulus control and sleep restriction in order to reverse maladaptive sleep habits (time in bed, napping, bedtime variability, rise time variability) proposed to maintain insomnia. It also involves the practice of sleep hygiene principles.
  Arms: Behavior Therapy
Behavioral: Waitlist. — The waitlist serves as a passive control which will receive the same measures administered to the cognitive and behaviour therapy groups.
  Arms: Waitlist

SUMMARY:
The overall purpose with this investigation is to further our knowledge about cognitive behavioral therapy (CBT) for insomnia by examining treatment components, mediators, and moderators. The first aim that will be addressed is to explore the efficacy of the CBT components with a dismantling-treatment strategy. Two active CBT interventions, intended to define its components - cognitive therapy and behavior therapy - will be compared with one another as well as with a waitlist condition on a broad range of outcomes at five to nine assessment points depending on the measures. The design will thus enable us to examine what CBT component or components are necessary, sufficient and facilitative of therapeutic change. The second aim that will be explored is to investigate what processes occur in CBT that may contribute to treatment outcome with a treatment-mediator strategy. To examine mediators for CBT, the following mediators will be assessed; Anxiety and Preoccupation about sleep Questionnaire (APSQ), Dysfunctional Beliefs and Attitudes about Sleep (DBAS), Sleep Associated Monitoring Index (SAMI), Sleep-Related Behavior Questionnaire (SRBQ), time in bed, napping, bedtime variability, and rise time variability. The hypothesis is that cognitive processes will mediate cognitive therapy outcomes, and that behavioral factors will have a mediating role for behavior therapy improvements. The third aim that will be addressed is to examine what patient characteristics does CBT depend on to be effective with a treatment-moderator strategy. To investigate moderators for CBT, the following moderators will be assessed; age, gender, occupational status, level of education, initial insomnia severity, dysfunction, medication use, chronic pain, psychiatric co-morbidity, medical co-morbidity, behavioral and cognitive processes used as mediators will also be employed as moderators.

ELIGIBILITY:
Inclusion Criteria:

* Presence of insomnia more than three nights per week and for more than three months.
* Insomnia despite adequate opportunity to sleep.
* Insomnia severity typical for insomnia disorder, i.e. 11 points or more on the Insomnia Severity Index (ISI).
* Nighttime insomnia symptoms, i.e., two points or more on at least one of the first three ISI questions.
* Daytime insomnia symptoms, i.e. two points or more on one or both of the ISI distress and impairment items (numbers 5 and 7).
* Clinical insomnia symptoms from sleep diaries concerning three nighttime symptoms (difficulties with sleep initiation, difficulties with sleep maintenance, and early morning awakenings), i.e., thirty minutes or more on average on one or more of the symptoms.
* No current or past CBT-I treatment within the past 5 years.
* Time and opportunity to participate in treatment for ten weeks.
* Time and opportunity to read approximately fifteen pages per week and execute homework assignments for ten weeks.
* Access to a computer, email and internet.

Exclusion Criteria:

* Severe depression, i.e., more than 30 points on MADRS-S.
* Suicidal risk, i.e., 4 points or more on item 9 on MADRS-S.
* A high intake of alcohol or caffeine,
* Insomnia due to shiftwork or other sleep-disturbing events (e.g., pregnancy, small children, or animals in the sleep environment).
* Participants with a history of psychotic or bipolar disorder.
* If a somatic condition is reported, it is required that it is relatively stable and/or that the candidate is receiving treatment for the condition.
* When a candidate fulfills criteria for a psychiatric or somatic condition, it is required that insomnia is the disorder currently most distressing and disabling or that the insomnia remains despite treatment for the comorbid condition.
* Participants with the following primary sleep disorders will be excluded via the Duke Structured Interview for Sleep Disorders (DSISD): sleep apnea, restless legs syndrome, periodic limb movement disorder, circadian rhythm disorder, and parasomnias.
* If sleep medication is used, it is required that the use has been relatively stable during three months.
* If Selective Serotonin Reuptake Inhibitors (SSRI) use is reported, it is required that the onset of the medication was at least three months prior to the telephone interview.
* Participants who regularly consume sleep-disturbing medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Changes on the insomnia severity index (ISI). | Pretreatment (week 0), during treatment (i.e., at week: 2, 4, 6, 8), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.

SECONDARY OUTCOMES:
Changes on the Work and Social Adjustment Scale (WSAS). | Pretreatment (week 0), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.
Changes in sleep onset latency (SOL). | Pretreatment (week 0), during treatment (week: 2, 4, 6, 8) and post-treatment (week 10).
Changes in wake time after sleep onset (WASO). | Pretreatment (week 0), during treatment (week: 2, 4, 6, 8) and post-treatment (week 10).
Changes in early morning awakenings (EMA). | Pretreatment (week 0), during treatment (week: 2, 4, 6, 8) and post-treatment (week 10).
Changes in total sleep time (TST). | Pretreatment (week 0), during treatment (week: 2, 4, 6, 8) and post-treatment (week 10).
Changes in Hospital Anxiety and Depression Scale (HADS) | Pretreatment (week 0), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.
Changes in nighttime symptoms, by using item 1 - 3 from the primary outcome measure. | Pretreatment (week 0), during treatment (week: 2, 4, 6, 8), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.
Changes in impairment, by using item 5 and 6 from the primary outcome measure. | Pretreatment (week 0), during treatment (week: 2, 4, 6, 8), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.
Changes in distress, by using item 4 and 7 from the primary outcome measure. | Pretreatment (week 0), during treatment (week: 2, 4, 6, 8), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.
Changes in Brunnsviken Brief Quality of life index (BBQ) | Pretreatment (week 0), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.

OTHER OUTCOMES:
Credibility Expectancy Questionnaire (CEQ ). | During the first treatment module.
Client Satisfaction Questionnaire (CSQ-8). | Post-treatment (week 10).
Activity and adherence with treatment protocol (self developed questionnaire assessing treatment activity and adherence relating to text, homework and therapist support). | Post-treatment (week 10).
Sick-leave and other concomitant treatment (self developed questionnaire). | Post-treatment (week 10).
Adverse events (questionnaire from a previous similar study). | Post-treatment (week 10).
Changes in physical activity (self developed questionnaire). | Pretreatment (week 0) and post-treatment (week 10).
Changes in Ford Insomnia Response To Stress Test (FIRST). | Pretreatment (week 0) and post-treatment (week 10) for the waitlist.
Changes in Daytime Insomnia Symptom Response Scale (DISRS) | Pretreatment (week 0) and post-treatment (week 10) for the waitlist.
Montgomery Åsberg Depression Rating Scale (MADRS). | Pretreatment (week 0).
Changes in suicide risk (Item 9 from the MADRS). | Pretreatment (week 0), post-treatment (week 10) and follow-up at 6, 12, and 18 month after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Jansson Fröjmark, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sunnhed R, Hesser H, Andersson G, Carlbring P, Lindner P, Harvey AG, Jansson-Frojmark M. Mediators of cognitive therapy and behavior therapy for insomnia disorder: A test of the processes in the cognitive model. J Consult Clin Psychol. 2022 Sep;90(9):696-708. doi: 10.1037/ccp0000756. Epub 2022 Sep 8. PMID 36074617
- [Derived] Blanken TF, Jansson-Frojmark M, Sunnhed R, Lancee J. Symptom-specific effects of cognitive therapy and behavior therapy for insomnia: A network intervention analysis. J Consult Clin Psychol. 2021 Apr;89(4):364-370. doi: 10.1037/ccp0000625. Epub 2021 Feb 25. PMID 33630618
- [Derived] Sunnhed R, Hesser H, Andersson G, Carlbring P, Morin CM, Harvey AG, Jansson-Frojmark M. Comparing internet-delivered cognitive therapy and behavior therapy with telephone support for insomnia disorder: a randomized controlled trial. Sleep. 2020 Feb 13;43(2):zsz245. doi: 10.1093/sleep/zsz245. PMID 31608389
- See also: Comparative Efficacy of Behavior Therapy, Cognitive Therapy, and Cognitive Behavior Therapy for Chronic Insomnia: A Randomized Controlled Trial — https://www.ncbi.nlm.nih.gov/pubmed/24865869